CLINICAL TRIAL: NCT02002390
Title: Efficacy and Safety of FTY720 for the Treatment of Acute Stroke
Brief Title: Efficacy and Safety of FTY720 for Acute Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Fu-Dong Shi, Head of Neurology Department, Tianjin Medical University General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB2013-054-02
Record Dates: First submitted 2013-11-24; First posted 2013-12-05 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Stroke; Vascular Accident; Cerebral Stroke; Ischemic Cerebrovascular Accident; Stroke, Acute
Keywords: Stroke,Fingolimod(FTY 720), treatment
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fingolimod (FTY720) group (Experimental): Drug: Fingolimod capsules will be administered as 0.5mg/day over a course of 3 consecutive days after stroke onset.
  Interventions: Drug: Fingolimod
- Control group (Placebo Comparator): Patients will receive usual care and drug use in hospital.
  Interventions: Drug: Fingolimod

INTERVENTIONS:
Drug: Fingolimod — A sphingosine-1-phosphate receptor regulator
  Other Names: FTY720

SUMMARY:
Stroke is one of the main severe disease of public health importance. Increasing evidence suggests that inflammatory mechanisms plays a significant role in stroke. So, immune targets are supposed to be an effective one. The sphingosine-1-phosphate receptor regulator Fingolimod(FTY720)is an effective immunology modulator which has been widely used in autoimmune disease and has been testified effective on stoke animal models.

DETAILED DESCRIPTION:
This study will enroll 87 stroke patients who have been diagnosed with stroke and meet the inclusion criteria.

After successfully meeting initial screening criteria, investigators will contact the family, explain the study, and send a consent form for their review.

After that, patients will be given 0.5mg/day oral fingolimod over a course of 3 consecutive days , then investigators will make a neurofunctional assessment before and 7days, 30 days and 90days after oral fingolimod. And Magnetic Resonance of the brain before, 7days, 14days and 90days after oral fingolimod. Furthermore 5ml intravenous blood for flow cytometry is also taken before and 1day,3days,7days after fingolimod use.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Clinical presentation of spontaneous intracerebral hemorrhage/ischemic stroke
* MRI/MRA scan compatible with spontaneous intracerebral hemorrhage/ ischemic stroke
* Time to fty720 treatment< 72 h from symptom onset
* Glasgow Coma Score >6 on initial presentation or improvement to a Glasgow Coma Score >6 within the time frame for enrollment.
* Primary supratentorial ICH of ≥5cc and <30cc
* TOAST: Large-artery atherosclerosis

Exclusion Criteria:

* Patients who will undergo surgical evacuation of intracerebral hemorrhage
* Inability to undergo neuroimaging with Magnetic Resonance
* Glasgow Coma Score < 6.
* Baseline modified Rankin Scale score >1
* Primary intraventricular hemorrhage ICH due to coagulopathy (PT > 15 s or International Normalized Ratio > 1.3, Partial Thromboplastin Time > 36) or trauma
* Thrombocytopenia: platelet count <100 000
* Clinically significant hepatic disease as demonstrated by history, clinical exam (ascites, varices), or laboratory findings (LFTs >2x normal, coagulopathy as described)
* Comorbid conditions likely to complicate therapy including but not limited to the following: a history of New York Heart Association class II, III, or IV Congestive Heart Failure; end-stage acquired immune deficiency syndrome
* Pregnancy
* Malignancy (history of or active)
* Bradyarrhythmia and Atrioventricular Block
* Concomitant use with antineoplastic,immunosuppressive or immune modulating therapies
* Macular Edema

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-10; Primary Completion 2014-10-01 (Actual); Study Completion 2014-10-01 (Actual)

PRIMARY OUTCOMES:
Clinical improvement | up to 90 days
  Neurofunctional assessment including NIHSS, modified Barthel Index, modified Rankin Scale,and Glasgow coma scale are used to describe the clinical improvement at baseline, 7days, 14days, 30days and 90days.

SECONDARY OUTCOMES:
Change in image | up to 90 days
  Outcomes are measured at baseline, 7 days, 14 days and 90 days after onset
Change in immunology function | up to 7 days
  Use the flow cytometry to measure the change at baseline, 1 day, 3 days, 7 days after drug use

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Dong Shi, MD,PhD, Principal Investigator — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Li HD, Li R, Kong Y, Zhang W, Qi C, Wang D, Hao H, Liu Q. Selective Sphingosine 1-Phosphate Receptor 1 Modulation Augments Thrombolysis of Low-Dose Tissue Plasminogen Activator Following Cerebrovascular Thrombosis. Front Immunol. 2022 May 27;13:801727. doi: 10.3389/fimmu.2022.801727. eCollection 2022. PMID 35720286
- [Derived] Zhu Z, Fu Y, Tian D, Sun N, Han W, Chang G, Dong Y, Xu X, Liu Q, Huang D, Shi FD. Combination of the Immune Modulator Fingolimod With Alteplase in Acute Ischemic Stroke: A Pilot Trial. Circulation. 2015 Sep 22;132(12):1104-1112. doi: 10.1161/CIRCULATIONAHA.115.016371. Epub 2015 Jul 22. PMID 26202811
- [Derived] Fu Y, Hao J, Zhang N, Ren L, Sun N, Li YJ, Yan Y, Huang D, Yu C, Shi FD. Fingolimod for the treatment of intracerebral hemorrhage: a 2-arm proof-of-concept study. JAMA Neurol. 2014 Sep;71(9):1092-101. doi: 10.1001/jamaneurol.2014.1065. PMID 25003359